CLINICAL TRIAL: NCT05920460
Title: Cognitive Behavioral Therapy for Insomnia and Depression Among Menopausal Women: A Randomized Control Trial
Brief Title: Cognitive Behavioral Therapy for Insomnia and Depression Among Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Loutfy, Ph.D., Lecturer of Nursing, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hashem2023
Record Dates: First submitted 2023-04-19; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Depression; Insomnia; Cognitive Behavioral Therapy; Menopausal Depression
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Cognitive Behavioral Therapy group received seven weekly face-to-face sleep group Cognitive Behavioral Therapy sessions lasting for 50-60 min. The Cognitive Behavioral Therapy program was developed by the research team after reviewing the literature and consulting with experts. Cognitive Behavioral Therapy was held in a lecture hall located in the PPFK branch office before individual counseling was initiated.
  Interventions: Behavioral: Cognitive Behavioral Therapy Program
- Control Group (No Intervention): The study participants of the control arm were interviewed separately and were given general health advice.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy Program — Brief description of the Cognitive Behavioral Therapy program is given below:
  * Session 1: Mutual understanding and rapprochement
  * Session 2: Sleep hygiene education
  * Session 3: Psychoeducation about stimulus control strategies; monitoring sleep environments, and identification of behavioral habits at bedtime, dysfunctional beliefs, and attitudes about sleep.
  * Session 4: Training on relaxation techniques
  * Session 5: Psycho education about depression
  * Session 6: Cognitive restructuring
  * Session 7: The terminating session
  Arms: Experimental Group

SUMMARY:
Considering physical and psychological problems that threaten women during the menopausal period, it seems that therapies that can help women cope with these problems, especially psychological ones, will be useful. The community mental health nurse is usually the first health professional whom women rely on to relieve their menopause symptoms. It is essential for the primary health care nurse to know how to properly approach women at this stage of their life and how to provide them the best and safe treatment. Because only limited interventional studies have been done to manage insomnia and depression among menopausal women in Egypt, the present study focused on reducing and insomnia and depression of menopausal women by using group Cognitive behavioral therapy. The current study aimed to examine the efficiency of group Cognitive Behavioral Therapy for insomnia and depression among menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women with depression (BDI-II score of 14-63)
* Women aged between 40 and 55 years old, menopausal (12 consecutive months without menses)
* Women are willing to provide written informed consent to participate in the study.
* Women who have the ability to read and write Arabic language.
* Women who report wake after sleep onset (wakefulness in the middle of the night after falling asleep) of an hour or more on ≥ 3 nights per week and met criteria for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (American Psychiatric Association, 2013) insomnia disorder with onset or exacerbation during the peri- or postmenopausal period per clinical interview with the researcher.
* Women who have a total score of >5 on the Pittsburgh Sleep Quality Index (PSQI), which indicates poor sleep, and a total score of >7 on the Insomnia Severity Index (ISI), which indicates insomnia.

Exclusion Criteria:

* Women who are currently under any type of psychotherapy or have a previous experience of Cognitive Behavioral Therapy.
* Women who have a history of neuropsychiatric illness, cancer, chemotherapy, and sudden stress in the previous 6 months (due to unfortunate events in the family) or have a severe or uncontrolled physical illness.
* Women who are clearly diagnosed as having sleep disorders or obstructive sleep apnea and had taken sleeping medications.
* Women who are on hormonal replacement therapy or cancer therapy or drugs such as tricyclic antidepressants, selective serotonin reuptake inhibitors, sedatives, and other hormones; and those who had undergone hysterectomy with oophorectomy.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The main aim focused on women at age of menopause.
Enrollment: 88 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
The effect of Cognitive Behavioral Therapy on Womens' insomnia symptom | 8 - 12 weeks
  the women who received the Cognitive Behavioral Therapy would exhibit a significantly change in insomnia symptom after the program compared to women in the control group.
  The Insomnia Severity Index (ISI; Morin et al., 2011), the ISI aims to assess the severity of insomnia over the past 2 weeks.
The effect of Cognitive Behavioral Therapy on Womens' depressive levels | 8 - 12 weeks
  the women who received the Cognitive Behavioral Therapy would exhibit a significantly change in depressive levels after the program compared to women in the control group.
  The Beck Depression Inventory, 2nd edition (BDI-II; Beck et al., 1996), BDI-II aims to assess the depressive symptoms. It is a 21-item self-report statements about how the person had been feeling in the last week. The BDI-II scores range from 0 to 63, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Correlation between studied variables before application of the intervention | 8 - 12 weeks
  Sleep quality index investigates the correlation significantly to insomnia severity index and beck depression inventory.
  The Pittsburgh Sleep Quality Index (PSQI) 1989, the PSQI is a self-completed questionnaire that assesses sleep quality over the previous month. The scale has 19-items, five of which should be answered by bed mates or roommates.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Beni-Suef University, Banī Suwayf, Other
  - Mansoura University, Al Mansurah

REFERENCES:
- [Derived] El-Monshed AH, Khonji LM, Altheeb M, Saad MTE, Elsheikh MA, Loutfy A, Ali AS, El-Gazar HE, Fayed SM, Zoromba MA. Does a program-based cognitive behavioral therapy affect insomnia and depression in menopausal women? A randomized controlled trial. Worldviews Evid Based Nurs. 2024 Apr;21(2):202-215. doi: 10.1111/wvn.12707. Epub 2024 Feb 8. PMID 38329153